CLINICAL TRIAL: NCT03048552
Title: Family Engagement, Cross-System Linkage to Substance Use Treatment for Juvenile Probationers -- Phase 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Katherine Elkington, Associate Professor of Clinical Psychology (in Psychiatry), New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 7108; R34DA039316 (NIH)
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Results first posted 2022-05-11 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Substance Use; Substance Abuse; Substance Use Disorders; Substance-Related Disorders; Substance Dependence; Substance Related Problem
Keywords: drug use; drug addiction; drug habituation; drug use disorders; organic mental disorders; substance-induced; substance abuse; substance addiction; substance dependence; substance use disorders
MeSH Terms: conditions — Substance-Related Disorders; Neurocognitive Disorders

STUDY DESIGN:
Intervention Model Description: This study is a randomized control trial. Caregiver-youth dyads are randomized to either the control (standard of care) or experimental (Family CONNECT) group based on the youth's probation officer (randomization occurs at the level of the youth's probation officer). If randomized to the control (standard of care) group, caregiver-youth dyads will work with their probation officer as usual to link to substance use services. If randomized to the experimental (Family CONNECT) group, caregiver-youth dyads will work with a linkage specialist to link to substance use services. Youth in both groups will be compared to a baseline stand of care collected during the pre-implementation period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): This arm is comprised of caregiver-youth dyads randomized to work with the youth's probation officer as usual to link youth to substance use services.
- Family CONNECT (Experimental): This arm is comprised of caregiver-youth dyads randomized to work with linkage specialists to link youth to substance use services.
  Interventions: Behavioral: Family CONNECT

INTERVENTIONS:
Behavioral: Family CONNECT — Linkage specialists, who are clinical social workers and embedded within the probation departments, will work with specifically caregiver-youth dyads in the Family CONNECT arm to link youth to substance use services.
  Arms: Family CONNECT

SUMMARY:
Developed from adapting and combining two evidence-based programs, Project CONNECT (a linkage-to-services program that targets barriers within the probation and substance abuse treatment systems) and TIES (a program that teaches family engagement skills to providers), Family CONNECT is a linkage-to-services program that targets both family and system-level factors to increase youth use of and retention in substance use services. Using Linkage Specialists embedded within probation departments, Family CONNECT will be implemented in two NYS probation departments. This proposed study will evaluate the impact of Family CONNECT on (1) youth referral from probation to substance abuse treatment, (2) youth and family engagement in substance abuse treatment, (3) youth enrollment/retention in substance abuse treatment, and (4) youth substance use and recidivism. Counts of youth referred, youth who start treatment, and youth retained in treatment will be obtained from the juvenile justice agency for 6-months pre-implementation of Family Connect (i.e. baseline) and during the implementation period of e-Connect; counts of youth recidivism will be obtained 6 months following the completion of Family Connect. This study will also identify family and probation organizational factors influencing Family CONNECT implementation in probation settings. 50 caregiver-youth dyads and up to 36 probation officers will be recruited as participants in the study. Caregiver-youth dyads will be evaluated at baseline, 2 and 6 months; probation officers at baseline, 6, 12, and 18 months; linkage specialists at baseline, 6, 12, and 18 months.

ELIGIBILITY:
Youth:

Inclusion Criteria

1. Between 10-18 years of age
2. English speaking
3. A caregiver who will participate in the study
4. MAYSI-2 score of ≥ 4 on any MAYSI-2 subscale; YASI mental health and substance use screen items; or other documented evidence of mental health or substance use problem
5. Currently on probation

Exclusion Criteria 1. Cognitively unable to complete the interview

Caregiver:

Inclusion criteria

1. Youth's legal guardian (or permission from legal guardian)
2. Youth who will participate
3. English speaking

Exclusion criteria:

1. Cognitively unable to complete the interview

Probation staff:

Inclusion criteria:

1. Currently employed at probation department

Exclusion criterion:

1. None

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine S Elkington, PhD, Principal Investigator — New York State Psychiatric Institute

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by study staff, following probation officer referral, between December 2015-May 2017 in two county probation agencies. Probation officers were randomized into either the treatment of SOC arm so that probation officers worked exclusively with either youth in the treatment or SOC arm to avoid cross-contamination across study arms.
Pre-assignment Details: Following recruitment, if the youth-caregiver dyad were working with a probation officer (PO) that was in the treatment arm, they were linked with the Linkage Specialist and began the intervention. If they were working with a PO who was in the control arm, they were linked to services in the usual way.
  Study completion occurred when dyads completed their 6 month survey, and were linked to treatment (experimental arm only)
Groups:
- Standard of Care - Youth: This arm is comprised of youth from caregiver-youth dyads randomized to work with the youth's probation officer as usual to link youth to substance use services.
- Family CONNECT - Youth: This arm is comprised of caregiver-youth dyads randomized to work with linkage specialists to link youth to substance use services.
  Family CONNECT: Linkage specialists, who are clinical social workers and embedded within the probation departments, will work with specifically caregiver-youth dyads in the Family CONNECT arm to link youth to substance use services.
- Standard of Care - Caregiver: This arm is comprised of caregivers from caregiver-youth dyads randomized to work with the youth's probation officer as usual to link youth to substance use services.
- Family CONNECT - Caregiver: This arm is comprised of caregivers from caregiver-youth dyads randomized to work with linkage specialists to link youth to substance use services.
  Family CONNECT: Linkage specialists, who are clinical social workers and embedded within the probation departments, will work with specifically caregiver-youth dyads in the Family CONNECT arm to link youth to substance use services.
Period: Overall Study
Arm/Group | Standard of Care - Youth | Family CONNECT - Youth | Standard of Care - Caregiver | Family CONNECT - Caregiver
Started | 4 | 18 | 4 | 15 (Fewer caregivers were enrolled in Family CONNECT arm than youth as 2 caregivers had multiple children in the Family CONNECT arm: one caregiver had n=2 children and 1 caregiver had n=3 children.)
Completed | 4 | 18 | 4 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Family CONNECT - Youth: This arm is comprised of youth from caregiver-youth dyads randomized to work with linkage specialists to link youth to substance use services.
  Family CONNECT: Linkage specialists, who are clinical social workers and embedded within the probation departments, will work with specifically caregiver-youth dyads in the Family CONNECT arm to link youth to substance use services.
- Total: Total of all reporting groups
Arm/Group | Standard of Care - Youth | Family CONNECT - Youth | Family Connect - Caregiver | Standard of Care - Caregiver | Total
Number analyzed (Participants) | 4 | 18 | 15 | 4 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 18 | 0 | 0 | 22
  Between 18 and 65 years | 0 | 0 | 14 | 4 | 18
  >=65 years | 0 | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (1) | 14.9 (1.1) | 46.2 (10.5) | 39.5 (8.6) | 15.1 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 12 | 4 | 25
  Male | 3 | 10 | 3 | 0 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 8 | 2 | 1 | 11
  Not Hispanic or Latino | 4 | 10 | 13 | 2 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 5 | 6 | 1 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 13 | 9 | 3 | 29
Region of Enrollment [Number; unit: participants]
  United States | 4 | 18 | 15 | 4 | 41
County [Count of Participants; unit: Participants] — Participants were recruited from two counties in the state in which the study took place. To retain confidentiality, counties are labeled as County 1 and County 2
  Participants
    County 1 | 4 | 14 | 11 | 0 | 29
    County 2 | 0 | 4 | 4 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Youth Enrolled in Substance Use Treatment
Description: Count of youth participants enrolled in substance use treatment based on self-report or administrative records
Time Frame: Two years (study implementation period)
Population: Youth on probation with identified substance use need
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care- YOUTH: This arm is comprised of caregiver-youth dyads working with the youth's probation officer (PO) who was randomly assigned to the SOC arm, to work with the PO as usual to link youth to substance use services.
- Family CONNECT- YOUTH: This arm is comprised of caregiver-youth dyads working with a probation officer (PO) randomized to the experimental arm. These dyads then worked with linkage specialists to link youth to substance use services.
  Family CONNECT: Linkage specialists, who are clinical social workers and embedded within the probation departments, will work with specifically caregiver-youth dyads in the Family CONNECT arm to link youth to substance use services.
Arm/Group | Standard of Care- YOUTH | Family CONNECT- YOUTH
Number analyzed (Participants) | 4 | 18
Participants
  Enrolled | 0 | 12
  Did not enroll | 4 | 6

2. Primary Outcome: Youth Enrolled in Any Behavioral Health Treatment
Description: Number of youth enrolled in any behavioral health treatment (incl. mental health and substance use) within the past 6 months
Time Frame: Two years (study implementation period)
Population: Youth on probation with identified substance use need
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care- YOUTH | Family CONNECT- YOUTH
Number analyzed (Participants) | 4 | 18
Participants
  Attended intake appointment | 2 | 15
  No intake | 2 | 3
Statistical Analysis 1: Comparison: Standard of Care- YOUTH vs Family CONNECT- YOUTH; Test type: Superiority; p = 0.148, Fisher Exact

3. Secondary Outcome: Youth Referred for Substance Use Treatment
Description: Number of youth referred to substance use treatment
Time Frame: Two years (study implementation period)
Population: Youth on probation with identified substance use need
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care- YOUTH | Family CONNECT- YOUTH
Number analyzed (Participants) | 4 | 18
Participants
  Referred | 0 | 17
  No referral | 4 | 1
Statistical Analysis 1: Comparison: Standard of Care- YOUTH vs Family CONNECT- YOUTH; Test type: Superiority; p < 0.01, Fisher Exact

4. Secondary Outcome: Youth Referred for Any Behavioral Health Treatment
Description: Number of youth who are referred to any behavioral health treatment
Time Frame: two years (implementation period)
Population: Youth on probation with identified substance use need
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care- YOUTH | Family CONNECT- YOUTH
Number analyzed (Participants) | 4 | 18
Participants
  Referred to Behavioral Health | 4 | 17
  No Referral | 0 | 1
Statistical Analysis 1: Comparison: Standard of Care- YOUTH vs Family CONNECT- YOUTH; Test type: Superiority; p = 0.818, Fisher Exact

5. Other Pre Specified Outcome: Youth Initiated Substance Use Treatment
Description: Number of youth who attended an additional substance use treatment appointment following intake.
Time Frame: Two years (study implementation period)
Population: Youth on probation with identified substance use need
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care- YOUTH: This arm is comprised of caregiver-youth dyads randomized to work with the youth's probation officer as usual to link youth to substance use services.
- Family CONNECT- YOUTH: This arm is comprised of caregiver-youth dyads randomized to work with linkage specialists to link youth to substance use services.
  Family CONNECT: Linkage specialists, who are clinical social workers and embedded within the probation departments, will work with specifically caregiver-youth dyads in the Family CONNECT arm to link youth to substance use services.
Arm/Group | Standard of Care- YOUTH | Family CONNECT- YOUTH
Number analyzed (Participants) | 4 | 18
Participants
  Did not initiate treatment | 4 | 10
  Initiated Treatment | 0 | 8

6. Other Pre Specified Outcome: Youth Initiated Any Behavioral Health Treatment
Description: Number of youth who attended an additional behavioral health treatment appointment following intake.
Time Frame: two years (study implementation period)
Population: Youth on probation with identified substance use need
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care- YOUTH | Family CONNECT- YOUTH
Number analyzed (Participants) | 4 | 18
Participants
  Initiated Treatment | 2 | 9
  Did not initiate treatment | 2 | 9
Statistical Analysis 1: Comparison: Standard of Care- YOUTH vs Family CONNECT- YOUTH; Test type: Superiority; p = 0.625, Fisher Exact

ADVERSE EVENTS:
Time Frame: 6 months for standard of car arm; between 6 and 13 months for treatment arm
Groups:
- Standard of Care- Youth: This arm is comprised of youths randomized to work with the youth's probation officer as usual to link youth to substance use services.
- Family CONNECT- Youth: This arm is comprised of youths randomized to work with linkage specialists to link youth to substance use services.
  Family CONNECT: Linkage specialists, who are clinical social workers and embedded within the probation departments, will work with specifically caregiver-youth dyads in the Family CONNECT arm to link youth to substance use services.
- Standard of Care- Caregivers: This arm is comprised of caregivers from caregiver-youth dyads randomized to work with the youth's probation officer as usual to link youth to substance use services.
- Family CONNECT- Caregivers: This arm is comprised of caregivers from caregiver-youth dyads randomized to work with linkage specialists to link youth to substance use services.
  Family CONNECT: Linkage specialists, who are clinical social workers and embedded within the probation departments, will work with specifically caregiver-youth dyads in the Family CONNECT arm to link youth to substance use services.
Arm/Group | Standard of Care- Youth | Family CONNECT- Youth | Standard of Care- Caregivers | Family CONNECT- Caregivers
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/18 | 0/4 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/18 | 0/4 | 0/15
Other Adverse Events (participants affected / at risk) | 0/4 | 0/18 | 0/4 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT03048552/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT03048552/ICF_001.pdf